CLINICAL TRIAL: NCT03109210
Title: Therapist-Directed VS Online Therapy for Insomnia Co-Occuring With Sleep Apnea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HS2989
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Insomnia, Primary; Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Care (No Intervention): Participants randomized to standard care will receive normal follow-up care with their health care provider. This will include routine assessment and adjustment of PAP therapy, and instruction in proper sleep hygiene.
- Intervention (Experimental): In addition to standard care procedures, participants randomized to the intervention arm will receive up to two sequential treatments. First, participants will receive Online Cognitive Behavioral Therapy (OCBT). Those who meet criteria for remission after this first treatment will continue through follow-up without further treatment. Those who do not will be randomized again to either extended OCBT, or Therapist-directed Cognitive Behavioral Therapy (TCBT).
  Interventions: Behavioral: Online Cognitive Behavioral Therapy (OCBT); Behavioral: Therapist-directed Cognitive Behavioral Therapy (TCBT)

INTERVENTIONS:
Behavioral: Online Cognitive Behavioral Therapy (OCBT) — Cognitive behavioral therapy delivered via commercial online software.
  Other Names: OCBT
  Arms: Intervention
Behavioral: Therapist-directed Cognitive Behavioral Therapy (TCBT) — Cognitive Behavioral Therapy delivered via traditional, in-person interaction with a licensed mental health professional.
  Other Names: TCBT
  Arms: Intervention

SUMMARY:
This two-site randomized clinical trial will investigate and compare three treatments for insomnia in patients who have been diagnosed with and treated for sleep apnea: online cognitive behavioral therapy (OCBT), therapist-directed cognitive behavioral therapy (TCBT), and standard clinical care. 384 patients will be recruited and will attend up to 15 visits over 10 months. Visits will include baseline assessment, treatment visits, and post-treatment follow-up visits. Visits will involve completion of questionnaires, meeting with therapists, and a physical exam.

DETAILED DESCRIPTION:
This dual-site randomized clinical trial will use a "SMART" design to test a stepped care model relative to standard positive airway pressure (PAP) therapy and determine if (1) augmentation of PAP therapy with online Cognitive Behavioral Therapy improves short-term outcomes of comorbid obstructive sleep apnea(OSA)/insomnia; and (2) providing a higher intensity 2nd-stage cognitive behavioral therapy (CBT) to patients who show sub-optimal short-term outcomes with OCBT+PAP improves short and longer-term outcomes. After completing baseline assessment, the 384 comorbid OSA\insomnia patients enrolled will be randomized to a 1st-stage therapy that includes usual care PAP + OCBT (n=288) or UC (usual care PAP + sleep hygiene education; n=96). Insomnia and OSA will be reassessed after 8 weeks. OCBT recipients who meet "remission" criteria will continue PAP but be offered no additional insomnia intervention and will complete study outcome measures again after an additional 8-weeks and at 3 and 6 month follow-ups. OCBT recipients classified as "unremitted" after 8 weeks of treatment will be re-randomized to a 2nd-stage treatment consisting of continued, expanded engagement in OCBT or a switch to therapist-directed CBT (TCBT). Those receiving the 2nd-stage intervention as well as the UC group will be reassessed after another 8 weeks and at 3- and 6-month follow-up time points.

ELIGIBILITY:
Inclusion Criteria:

To be included participants must > 21 years old and:

1. have a diagnosis of OSA with an AHI > 5 on a diagnostic polysomnogram;
2. accept PAP as primary/sole OSA therapy, been given a prescription for PAP and filled it within the last 3 months, have had an opportunity to use PAP for at least one month, and show mean use of > 1 hour per night;
3. have a complaint of persistent (i.e., > 3 months) sleep onset or sleep maintenance difficulties despite having adequate opportunity for sleep and accompanied by significant daytime impairment or distress about poor sleep;
4. an Insomnia Severity Index (ISI) score > 10 indicating at least "mild" insomnia; and
5. a sleep onset latency or wake time after sleep onset > 30 minutes 3 or more nights per week during two weeks of sleep diary monitoring.

Exclusion Criteria:

1. an untreated psychiatric disorder (e.g., major depression) found on structured interviews as these conditions have specific treatments and it would be inappropriate not to offer those treatments;
2. a lifetime diagnosis of any psychotic or bipolar disorder as sleep restriction for insomnia may precipitate hallucinations and mania;
3. an imminent risk for suicide;
4. alcohol or drug abuse within the past year;
5. terminal illness (e.g., cancer), or neurological degenerative disease (e.g., dementia);
6. current use of medications known to cause insomnia (e.g., stimulants);
7. comorbid narcolepsy, idiopathic hypersomnia, restless legs syndrome (score of >11 in the IRLS), periodic limb movement during sleep (known PLMS with arousal > 15 per hour), or a circadian rhythm sleep disorder if habitual bedtimes are later than 3:00 AM or rising times are later than 11:00 AM; or
8. consuming > 2 alcoholic beverages per day on a regular basis; or
9. consuming more than 10 caffeinated beverages per day on a regular basis; or
10. consuming marijuana in any form on a regular basis >1 time per week, or if used after 4:00 p.m; or
11. change in thyroid medication dosage or received a new prescription for thyroid medication 3 months before the screening visit; or
12. physician-diagnosed or self-reported seizure disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) score change | Symptom remission will be measured at post-treatment visits one and two, approximately 18 and 28 weeks following enrollment.
  Change in participants' score on the ISI will be measured over baseline, post-treatment, and follow-up visits.
Quebec Sleep Questionnaire (QSQ) score change | Participants will be asked to complete the QSQ at baseline, post-treatment, and follow-up visits, at approximately weeks 1, 18, and 28.
  Change in participants' score on the QSQ will be measured over baseline, post-treatment, and follow-up visits.

SECONDARY OUTCOMES:
Change in subjective measurement of total sleep time | Participants will be asked to complete two weeks of sleep diaries at baseline (week 1), post-treatment (weeks 8 and 18), and follow-up visits (months 9 and 12) to measure change in these assessments over time.
  Participants will be asked to fill out a sleep diary throughout the study. Study personnel will use these diaries to calculate subjective assessment of total sleep time.
Change in subjective measurement of sleep efficiency | Participants will be asked to complete two weeks of sleep diaries at baseline (week 1), post-treatment (weeks 8 and 18), and follow-up visits (months 9 and 12) to measure change in these assessments over time.
  Participants will be asked to fill out a sleep diary throughout the study. Study personnel will use these diaries to calculate subjective assessment of sleep efficiency.
Positive Airway Pressure (PAP) Therapy Adherence | Adherence data will be collected through study completion, an average of one year.
  Participants' adherence to PAP therapy will be passively monitored during their participation in the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford Univeristy, Palo Alto, California
  - National Jewish Health, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eldridge-Smith ED, Manber R, Tsai S, Kushida C, Simmons B, Johnson R, Horberg R, Depew A, Abraibesh A, Simpson N, Strand M, Espie CA, Edinger JD. Stepped care management of insomnia co-occurring with sleep apnea: the AIR study protocol. Trials. 2022 Sep 24;23(1):806. doi: 10.1186/s13063-022-06753-4. PMID 36153634